CLINICAL TRIAL: NCT01527097
Title: Atorvastatin to Reduce Psoriasis Severity and Improve Endothelial Function in Patients With Severe Psoriasis and Non-Elevated LDL Levels: A Randomized, Double Blind, Placebo-Controlled Study.
Brief Title: Influence of Atorvastatin on Psoriasis Severity and Endothelial Function
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: We strongly feel that the ability to recruit the required number of patients is very low and thus decided to stop the study.
Sponsor: shmuel fuchs (Other)
Responsible Party: Sponsor-Investigator, shmuel fuchs, Prof Shmuel Fuchs, MD, MACC, FSCAI, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0263 - 11 - RMC
Record Dates: First submitted 2012-01-15; First posted 2012-02-06 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Psoriasis
Keywords: Cardiovascular Diseases; Pharmacologic Actions; Endothelial Function; Dermatology; Inflammatory Disease; Skin Disease
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases; Skin Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental)
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Atorvastatin placebo

INTERVENTIONS:
Drug: Atorvastatin — Drug: Atorvastatin 80 mg for 6 months following by 40 mg for additional 6 months once daily.
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Atorvastatin placebo — Atorvastatin 80mg during 6 month and 40mg in additional 6 month period once daily.
  Arms: Placebo

SUMMARY:
Patients with psoriasis seem to have increased risk for developing atherosclerosis. This may be due to the fact that psoriasis and atherosclerosis are both caused by inflammation and involvement of cells of the immune system. Atherosclerosis is frequently treated by statins (class of cholesterol lowering drugs), which lower bad cholesterol levels and also reduce inflammation. Some new evidences also suggest that therapy with statins may improve psoriasis skin disease.

The current study aims are to evaluate whether a strong statin named Atorvastatin can improve psoriatic skin disease and functioning of the arteries. The study also aims to evaluate if the activity of these two diseases are related to levels of common inflammatory biomarkers (substance in blood) and whether Atorvastatin can change their levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* Patients with psoriasis of at least 3-years duration
* Current moderate to severe psoriatic disease (PASI ≥12, IGA≥3)
* Statin-naïve patients
* No history of cardiovascular disease (ischemic heart disease, peripheral vascular disease or cerebrovascular disease)
* LDL levels

  * LDL level > 70 mg% and < 160 mg% in low risk patients (defined as having none or a single risk factor*)
  * LDL > 70 mg% and < 130 mg% in moderate risk patients (defined as the presence of 2 or more risk factors*)
  * LDL > 70 mg% and < 100 mg% in patients with type II diabetes
* hsCRP ≥ 1 mg/l * Risk factors: smoking, hypertension (blood pressure > 140/90 or current treatment with blood pressure lowering agents, HDL < 40 mg%, family history of premature coronary artery disease in a first degree relative younger than 45 (men) or 55 (women) and obesity (BMI ≥ 30).

Exclusion Criteria:

* Current statin therapy
* Patents with Atrial Fibrillation
* Elevated liver enzymes (> X3 ULN)
* History of statin-induced liver enzyme elevation
* Elevated CPK levels (> X3 ULN)
* History of myopathy including statin-induced
* Severe chronic renal failure (GFR <30 ml/min)
* Pregnant or breast-feeding women
* Individuals at risk for poor protocol, or medication compliance
* Patients with life-expectancy of less than 2 years
* Patients who are currently participating in another clinical trial
* Other current active inflammatory and/or infectious conditions
* Sensitivity to any of atorvastatin ingredients
* Concomitant drug therapy, taken on a regular basis, which may interact with Atorvastatin

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome variable of the study is defined as the composite endpoint of improving of psoriatic severity and endothelial function (assessed by FMD changes). | 3,6 and 12 months after randomization.
  Patient invited to clinic visits at 3,6 and 12 month follow up.At this visits in addition primary outcome will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Fuchs, Professor, Study Director — Rabin Medical Center, Israel
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel